CLINICAL TRIAL: NCT06005142
Title: Therapeutic Intervention of Nutraceutical Eriomin Associated with Metformin to Improve the Control of Hyperglycemia in Patients with Prediabetes: a Double-blind, Randomized, Placebo-controlled Crossover Clinical Trial
Brief Title: Therapeutic Intervention of Eriomin Associated with Metformin in the Control of Hyperglycemia in Pre-Diabetic Patients
Acronym: Eriomin+Met
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Thais Cesar (Other)
Collaborators: Ingredients by Nature TM (Unknown)
Responsible Party: Sponsor-Investigator, Thais Cesar, Visiting Professor, São Paulo State University
Organization: São Paulo State University (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SaoPSU23
Record Dates: First submitted 2023-03-27; First posted 2023-08-22 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Pre-diabetes
Keywords: citrus flavonoids; Eriomin; oral antidiabetic biguanide (metformin); hyperglycemia; microbiota
MeSH Terms: conditions — Glucose Intolerance; Hyperglycemia | interventions — WASH protein, Drosophila

STUDY DESIGN:
Intervention Model Description: A crossover, randomized, placebo-controlled, double-blind clinical trial will be conducted for 12 weeks, with a two-week washout interval, followed by another 12 weeks, totaling 26 weeks.
  All participants must be under oral biguanide (metformin) (1000 mg/day) regimen by at least two weeks before the intervention, and they will be measure for glycemia, HbA1c and OGTT, and an interview with an MD and Nutritionist in order to confirm eligibility, according to the inclusion/exclusion criteria.
  The selected individuals will be randomly distributed into 2 groups, and they will receive alternately Eriomin (or placebo), followed by 2-weeks of washout, and placebo (or Eriomin) for 12 weeks.
  At the beginning of the first, 12th, 14th, and 26th weeks, all subjects will be evaluated for the following: Glycemia, OGTT, HbA1c, Insulin, Lipids, TEAC, MDA, GLP-1, inflammatory, hepatic, kidney, and anthropometric parameters, and microbiota composition.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All subjects and the principal investigator will remain blinded to treatment until data analysis is complete. Eriomin (lemon flavonoids extract) and Placebo (composed of microcrystalline corn starch) were encapsulated in tablets of the same size, shape, and color, by a registered pharmacist.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Eriomin/Placebo (Active Comparator): Group A will receive Eriomin (250 mg/day) for 12 weeks, followed by a 2-week washout period, and then placebo (250 mg/day) for 12 weeks.
  Interventions: Dietary Supplement: Eriomin; Dietary Supplement: Washout; Dietary Supplement: Placebo
- Placebo/Eriomin (Placebo Comparator): Group B will receive placebo (250 mg/day) for 12 weeks, followed by a 2-week washout period, and then Eriomin (250 mg/day) for 12 weeks.
  Interventions: Dietary Supplement: Eriomin; Dietary Supplement: Washout; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Eriomin — Pre-diabetic patients on oral biguanide (metformin) (1000 mg/day) will receive a 250 mg/day capsule of Eriomin for 12 weeks.
Dietary Supplement: Washout — After 12 weeks of treatment with the active component (Eriomin) or placebo, the participants will follow a washout for 2 weeks.
Dietary Supplement: Placebo — Pre-diabetic patients on oral biguanide (metformin) (1000 mg/day) will receive a 250 mg/day placebo capsule for 12 weeks.

SUMMARY:
Citrus bioflavonoids, such as eriocitrin, hesperidin and naringin, have been shown improved hyperglycemia, insulin resistance and systemic inflammation, related to the development of type 2 diabetes. The nutraceutical Eriomin, a lemon flavonoid extract composed mainly by eriocitrin (70%) and other flavonoids (30%), improved the control of moderate hyperglycemia in pre-diabetic and diabetic patients without drug therapy. However, most patients with pre-diabetes are on oral biguanide (metformin) therapy, despite its limited efficacy (30-40%) on glycemic control and its undesirable gastrointestinal effects.

Therefore, in the current study, Eriomin will be administered at a dose of 250 mg/d to adults diagnosed with pre-diabetes and being treated with metformin (1,000 mg/d). This clinical trial was designed as a placebo-control, double-blind, two-arm, crossover design. Clinical characteristics, body composition, food consumption, metabolic and inflammatory biomarkers and the microbiota of all patients will be evaluated before, during and at the end of the 12-week period (arm). Biochemical and metabolic parameters associated with prediabetes are expected to improve or return to normal with Eriomin in combination with metformin. At the same time, an increase in beneficial intestinal bacteria is expected, reducing pre-diabetic dysbiosis, and perhaps a noticeable improvement in body composition.

DETAILED DESCRIPTION:
Recent evidence shows that bioflavonoids from citrus fruits and herbs can reduce hyperglycemia, dyslipidemia, insulin resistance and the systemic inflammatory process related to type 2 diabetes (T2D). Although they can be found in fruits and herbs, bioflavonoid supplements and nutraceuticals can provide sufficient and safe amounts of bioactive compounds to prevent the development of metabolic disorders, such as metabolic syndrome, diabetes, obesity and others. Eriocitrin flavanone, present in lemons, limes and oranges, has demonstrated anti-inflammatory, anti-hyperglycemic and antioxidant properties and is an integral part of lemon bioflavonoid supplements that have been widely marketed.

Eriocitrin metabolism, similar to hesperidin, is resistant to pancreatic enzymes and are mostly deglycosylated by intestinal bacteria (Bacteroides distasonis or Bacteroides uniformis) to eriodictyol before absorption. A minimal amount can be absorbed as glycosylated in the upper intestine. Eriodictyol, the aglycon of eriocitrin, can be metabolized by intestinal bacteria (with 3,4-dihydroxycinnamic acid formation) to homoeriodictyol and hesperetin through methoxylation. In the liver, eriodictyol is metabolized into glucuronides and conjugated sulfates of eriodictyol, homoeriodictyol, and hesperitin, through sulfation, glucuronidation and methylation, and later released into the circulation to exert biological activity.

Eriocitrin can increase the total antioxidant capacity, leading to a decrease in inflammatory markers (IL-6, MCP-1 and us-CRP) in the blood and organs of mice supplemented with the flavonoid. Eriocitrin also increased catalase and glutathione enzymes in the liver of diabetic rats, and decreased lipid peroxidation in blood, liver and kidney. Furthermore, oral administration of eriodictyol to diabetic rats improved glucose metabolism in the blood, liver and kidney, and suppressed diabetes by upregulating PPARγ29 mRNA expression.

Based on this experimental evidence, the nutraceutical Eriomin, composed of lemon bioflavonoids, was tested as a dietary supplement to control mild to moderate hyperglycemia in pre-diabetic and diabetic patients. After three months of therapy, there was a decrease in hyperglycemia, improvement in insulin resistance and a decrease in HbA1c.

Thus, the hypothesis of the current study is to use the nutraceutical Eriomin as a co-adjuvant to oral biguanide (metformin) therapy, improving control of hyperglycemia and insulin resistance, while increasing efficacy with a low dosage (250 mg/d) of the nutraceutical. It is expected to improve the quality of the microbiota, the glucose metabolism and body composition, in addition to reducing the side effects associated with the continuous use of metformin.

Therefore, the main objective of this study is to evaluate the effects of Eriomin (250mg/day) associated with metformin on glycemic control, insulin resistance and other metabolic, inflammatory and clinical parameters. Furthermore, it will evaluate changes in the microbiota of pre-diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Glycemia of 6.1 to 7.0 mmol / L
* Glycated hemoglobin with values between 5.7 and 6.4%

Exclusion Criteria:

* use of drugs, vitamins and dietary supplements, alcohol consumption (> 20 g alcohol/d), and intense physical activity (> 5 hours/week).
* History of cardiovascular disease, diabetes mellitus, liver, kidney or pancreatic disease

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Fasting Glycemia | 0-12-18-26 week
  Dosages of glycemia concentration (mg/dL) before and after intervention with Eriomin/placebo

SECONDARY OUTCOMES:
Oral Glucose Tolerance Test (OGTT) | 0-12-18-26 week
  Changes in blood glucose 2 hours after the oral glucose tolerance test (mg/dL) before and after intervention with Eriomin/placebo
HbA1c | 0-12-18-26 week
  Dosages of glycated hemoglobin (%) in the blood serum/plasma before and after intervention with Eriomin/placebo
Insulin | 0-12-18-26 week
  Dosages of Insulin (µU/mL) in the blood serum/plasma before and after intervention with Eriomin/placebo
Blood Lipids profile | 0-12-18-26 week
  Dosages of cholesterol (mg/dL), HDL-cholesterol (mg/dL) and triglycerides (mg/dL) in the blood serum/plasma before and after intervention with Eriomin/placebo
Antioxidant Capacity | 0-12-18-26 week
  Dosages of Trolox equivalent antioxidant capacity (TEAC) (μM) in the blood serum/plasma before and after intervention with Eriomin/placebo
Lipid Peroxidation | 0-12-18-26 week
  Dosages of Malondialdehyde (MDA) (mM) the blood serum/plasma before and after intervention with Eriomin/placebo
Glucagon-like peptide-1 (GLP-1) | 0-12-18-26 week
  Dosages of GLP-1 (pmol/L) the blood serum/plasma before and after intervention with Eriomin/placebo
Inflammatory parameters | 0-12-18-26 week
  Dosages of C Reactive Protein (CRP) (mg/dL), TNF-alpha (mg/dL), IL-6 (mg/dL) in the blood serum/plasma before and after intervention with Eriomin/placebo
Hepatic Enzymes | 0-12-18-26 week
  dosages of alkaline phosphatase (U/L), gamma glutamyl transferase (U/L), aspartate aminotransferase (U/L), and alanine aminotransferase (U/L) in the blood serum/plasma before and after intervention with Eriomin/placebo
Kidney Blood Parameters | 0-12-18-26 week
  Dosages of urea (mg/dL) and creatinine (mg/dL) in the blood serum/plasma before and after intervention with Eriomin/placebo
Anthropometric Parameters | 0-12-18-26 week
  Measurements of body weight (kg), muscle mass (kg), fat mass (kg) before and after intervention with Eriomin/placebo
Microbiota composition by 16S rRNA gene sequencing | 0-12-18-26 week
  Dosages of the main bacteria groups by Operational Taxonomic Units (OTU) and % of relative abundance by group

CONTACTS AND LOCATIONS:
Overall Officials: Thais B Cesar, PhD, Principal Investigator — São Paulo State University; Maria Rita M De Oliveira, PhD, Study Director — São Paulo State University; Valeria Cristina Samdrim, PhD, Study Chair — São Paulo State University; Katia Sivieri, PhD, Study Chair — São Paulo State University; Adriana Lucia Mendes, PhD, Study Chair — São Paulo State University; Gabriela A Meira, Nutrition, Study Chair — São Paulo State University
Locations (1):
- Centro de Estudos e Praticas em Nutrição (CEPRAN), Botucatú, São Paulo, Brazil

REFERENCES:
- [Background] Testa R, Bonfigli AR, Genovese S, De Nigris V, Ceriello A. The Possible Role of Flavonoids in the Prevention of Diabetic Complications. Nutrients. 2016 May 20;8(5):310. doi: 10.3390/nu8050310. PMID 27213445
- [Background] Vinayagam R, Xu B. Antidiabetic properties of dietary flavonoids: a cellular mechanism review. Nutr Metab (Lond). 2015 Dec 23;12:60. doi: 10.1186/s12986-015-0057-7. eCollection 2015. PMID 26705405
- [Background] Minato K, Miyake Y, Fukumoto S, Yamamoto K, Kato Y, Shimomura Y, Osawa T. Lemon flavonoid, eriocitrin, suppresses exercise-induced oxidative damage in rat liver. Life Sci. 2003 Feb 21;72(14):1609-16. doi: 10.1016/s0024-3205(02)02443-8. PMID 12551749
- [Background] Hiramitsu M, Shimada Y, Kuroyanagi J, Inoue T, Katagiri T, Zang L, Nishimura Y, Nishimura N, Tanaka T. Eriocitrin ameliorates diet-induced hepatic steatosis with activation of mitochondrial biogenesis. Sci Rep. 2014 Jan 15;4:3708. doi: 10.1038/srep03708. PMID 24424211
- [Background] Miyake Y, Shimoi K, Kumazawa S, Yamamoto K, Kinae N, Osawa T. Identification and antioxidant activity of flavonoid metabolites in plasma and urine of eriocitrin-treated rats. J Agric Food Chem. 2000 Aug;48(8):3217-24. doi: 10.1021/jf990994g. PMID 10956094
- [Background] Ferreira PS, Spolidorio LC, Manthey JA, Cesar TB. Citrus flavanones prevent systemic inflammation and ameliorate oxidative stress in C57BL/6J mice fed high-fat diet. Food Funct. 2016 Jun 15;7(6):2675-81. doi: 10.1039/c5fo01541c. Epub 2016 May 16. PMID 27182608
- [Background] Ribeiro CB, Ramos FM, Manthey JA, Cesar TB. Effectiveness of Eriomin(R) in managing hyperglycemia and reversal of prediabetes condition: A double-blind, randomized, controlled study. Phytother Res. 2019 Jul;33(7):1921-1933. doi: 10.1002/ptr.6386. Epub 2019 Jun 11. PMID 31183921
- [Background] Cesar TB, Ramos FMM, Ribeiro CB. Nutraceutical Eriocitrin (Eriomin) Reduces Hyperglycemia by Increasing Glucagon-Like Peptide 1 and Downregulates Systemic Inflammation: A Crossover-Randomized Clinical Trial. J Med Food. 2022 Nov;25(11):1050-1058. doi: 10.1089/jmf.2021.0181. Epub 2022 Jul 7. PMID 35796695
- [Background] Flory J, Lipska K. Metformin in 2019. JAMA. 2019 May 21;321(19):1926-1927. doi: 10.1001/jama.2019.3805. PMID 31009043
- [Derived] Cesar T, Oliveira MR, Sandrim V, Mendes A, Bruder R, Oliveira R, Sivieri K, Milenkovic D. Citrus flavonoid supplement enhances glycemic and metabolic control in prediabetic patients on metformin: a randomized controlled trial. Front Nutr. 2025 Aug 19;12:1639901. doi: 10.3389/fnut.2025.1639901. eCollection 2025. PMID 40904779